CLINICAL TRIAL: NCT00986245
Title: An Open-label, Multi-center, Crossover Study to Compare the Effect of Once-daily Ropinirole PR and Twice-daily Ropinirole PR in Patients With Parkinson Disease
Brief Title: Study to Compare the Effect of Ropinirole Prolonged Release Once-daily Versus Twice-daily
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0908-037-290
Record Dates: First submitted 2009-09-24; First posted 2009-09-29 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Ropinirole
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropinirole PR QD first, then BID (Active Comparator): Give Roipinirole prolonged release (PR) once-daily (QD) dose first, then twice-daily (BID) dosing
  Interventions: Drug: Ropinirole Prolonged release
- Ropinirole PR BID first, and then QD (Active Comparator): Give Ropinirole prolonged release (PR) twice-daily (BID) dosing, and then once-daily (QD) dosing
  Interventions: Drug: Ropinirole Prolonged release

INTERVENTIONS:
Drug: Ropinirole Prolonged release — Change Ropinirole immediate release or Pramipexole immediate release to Ropinirole prolonged release (PR) once-daily or twice-daily
  Other Names: Requip PD®

SUMMARY:
1. In order to compare the benefit, side effects, and patient preference of Ropinirole prolonged release when used in once-daily or twice-daily dosing
2. In order to estimate the conversion rate of dopamine agonists into Ropinirole prolonged release

DETAILED DESCRIPTION:
1. Study subjects : Parkinson disease who are on Ropinirole immediate release or Pramipexole immediate release and are considering to change into Ropinirole prolonged release
2. Cross over study design:

   * Group 1: once daily dose for 2 month then into twice daily in divided dose for 2 months
   * Group 2: twice daily in divided dose for 2 months then into once daily dose for 2 months
3. Dose adjustment may be done in the first 4 weeks.
4. Compare the benefit,side effects, and patient preference between the once daily vs twice daily dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-80
2. Parkinson disease
3. On dopamine agonists (Ropinirole IR or Pramipexole IR) and are considering to change into Ropinirole PR
4. On stable antiparkinsonian medication for at least 4 weeks
5. Who signed consent to the study

Exclusion Criteria:

1. Who are on less than 2 mg of Ropinirole IR or 0.375 mg of Pramipexole IR
2. Who have dementia, psychosis, major depression and other serious neurological or medical problems
3. Who are allergic to the similar medications
4. Who has history of heavy metal poisoning
5. Who were on othe clinical trials of other medications within the last 4 weeks
6. Whoa re pregnant or lactating
7. Who are considered not eligible by the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Boramae City Hospital, Seoul

REFERENCES:
- [Background] Lyons KE, Pahwa R. An open-label conversion study of pramipexole to ropinirole prolonged release in Parkinson's disease. Mov Disord. 2009 Oct 30;24(14):2121-7. doi: 10.1002/mds.22750. PMID 19768728
- [Background] Stocchi F, Hersh BP, Scott BL, Nausieda PA, Giorgi L; Ease-PD Monotherapy Study Investigators. Ropinirole 24-hour prolonged release and ropinirole immediate release in early Parkinson's disease: a randomized, double-blind, non-inferiority crossover study. Curr Med Res Opin. 2008 Oct;24(10):2883-95. doi: 10.1185/03007990802387130. Epub 2008 Sep 2. PMID 18768106
- [Derived] Yun JY, Kim HJ, Lee JY, Kim YE, Kim JS, Kim JM, Jeon BS. Comparison of once-daily versus twice-daily combination of ropinirole prolonged release in Parkinson's disease. BMC Neurol. 2013 Sep 2;13:113. doi: 10.1186/1471-2377-13-113. PMID 24004540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled in September 2009 and the last subject completed the study in December 2010.
Pre-assignment Details: A total of 82 patients with PD were enrolled in this study at two centers in Seoul, Korea.
Groups:
- Ropinirole PR-Once Daily First, Then Twice Daily: Ropinirole prolonged release(PR) once daily in first intervention period and twice daily in second intervention period (without washout period)
- Ropinirole PR-Twice Daily First, Then Once Daily: Ropinirole prolonged release(PR) twice daily in first intervention period and once daily in second intervention period (without washout period)
Period: First Intervention
Arm/Group | Ropinirole PR-Once Daily First, Then Twice Daily | Ropinirole PR-Twice Daily First, Then Once Daily
Started | 41 | 41
Completed | 31 | 33
Not Completed | 10 | 8
Not completed — Poor compliance | 8 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Out of indication | 1 | 0
Period: Second Intervention
Arm/Group | Ropinirole PR-Once Daily First, Then Twice Daily | Ropinirole PR-Twice Daily First, Then Once Daily
Started | 31 | 33
Completed | 29 | 32
Not Completed | 2 | 1
Not completed — Poor compliance | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive once daily first and twice daily first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 32
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 82

OUTCOME MEASURES:

1. Primary Outcome: Patient Preference
Description: Patient preference between once-daily and twice-daily regimen
Time Frame: After 16 weeks or at last visit for early completion
Population: Primary outcome measure was the preference of the subjects between once-daily versus twice-daily of RPR at the completion or at early completion after crossover.
  61 of participants completing period with study intervention.
Measure: Number; unit: participants
Groups:
- Once-daily: Once-daily preferred group
- Twice-daily: Twice-daily preferred group
- No Preference: No preference group
Arm/Group | Once-daily | Twice-daily | No Preference
Number analyzed (Participants) | 61 | 61 | 61
participants | 17 | 31 | 13

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale, Part 3
Description: Unified Parkinson's disease rating scale (UPDRS) motor scale after 8 weeks in each arm or at last visit for early completion.
  UPDRS part 3 is motor scale for parkinson's disease. Range: 0~108 Higher values represent more severe motor symptoms of parkinsonism.
Time Frame: 8 weeks for each arm or at last visit
Population: Total number of patients are 61 (Group 1 + Group 2), because of Crossover design. Once-daily or Twice-daily arm means clinical variables measured in once-daily or twice-daily regimen, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Once-daily of Ropinirole PR: Once-daily regimen of Ropinirole Prolonged release administered in either first intervention peirod or second intervention period.
- Twice-daily of Ropinirole PR: Twice-daily regimen of Ropinirole Prolonged release administered in either first intervention peirod or second intervention period.
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
units on a scale | 17.5 (8.2) | 17.1 (8.9)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; The UPDRS-part3 was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Non-Inferiority or Equivalence — 80% power; p < 0.05, Sign test; Mean Difference (Net) = 0.4

3. Secondary Outcome: Hoehn and Yahr Stage
Description: Hoehn and Yahr(HY) stage for parkinsonism after 8 weeks in each arm or at last visit for early completion Range: 0~5 Higher values represent more severe parkinsonism
Time Frame: 8 weeks for each arm or at last visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Once-daily of Ropinirole PR: Once-daily regimen of Ropinirole PR administered in either first intervention peirod or second intervention period.
- Twice-daily of Ropinirole PR: Twice-daily regimen of Ropinirole PR administered in either first intervention peirod or second intervention period.
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
Scores on a scale | 2.1 (0.5) | 2.1 (0.6)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; The Hoehn and Yahr stage was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Non-Inferiority or Equivalence — 80% power; p < 0.05, Sign test; Mean Difference (Net) = 0.0

4. Secondary Outcome: Overall Quality of Sleep
Description: Sleep questionnaire 1 for "Overall quality of sleep" Visual analogue scale: 0~10 Higher values represent worse overall sleep quality.
Time Frame: 8 weeks for each arm or at last visit
Population: Total number of patients are 61 (Group 1 + Group 2), because of Crossover design. QD or BID arm means clinical variables measured in once-daily or twice-daily regimen, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
units on a scale | 2.9 (2.6) | 3.2 (2.5)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; The "Overall quality of sleep" was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Non-Inferiority or Equivalence — 80% power; p < 0.05, Sign test; Mean Difference (Net) = 0.3

5. Secondary Outcome: Nocturnal Off-symptoms
Description: Sleep questionnaire 2 for "Nocturnal off-symptoms" Visual analogue scale: 0~10 Higher values represent worse nocturnal off-symptoms.
Time Frame: 8 weeks for each arm or at last visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
units on a scale | 2.9 (3.2) | 3.1 (3.2)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; The "Nocturnal off-symptoms" was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Non-Inferiority or Equivalence — 80% power; p < 0.05, Sign test; Mean Difference (Net) = 0.2

6. Secondary Outcome: Early Morning Off Symptoms
Description: Sleep questionnaire 3 for "early morning off symptoms" Visual analogue scale: 0~10 Higher values represent worse early morning off symptoms.
Time Frame: 8 weeks for each arm or at last visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
units on a scale | 2.5 (3.3) | 2.9 (3.2)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR; The "Early morning off symptoms" was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Superiority or Other; p < 0.05, Sign test — 80% power; Mean Difference (Net) = 0.4

7. Secondary Outcome: Epworth Sleep Scale
Description: Epworth sleep scale after 8 weeks in each arm or at last visit for early completion.
  Range: 0~24 Higher values represent worse daytime-sleepiness.
Time Frame: 8 weeks in each arm or at last visit for early completion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
units on a scale | 6.3 (5.2) | 6.4 (4.8)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; The "Epworth sleep scale" was compared between the Once-daily of Ropinirole PR arm and the Twice-daily of Ropinirole PR using the Wilcoxon signed rank test; Test type: Non-Inferiority or Equivalence — 80% power; p < 0.05, Sign test; Mean Difference (Final Values) = 0.1

8. Secondary Outcome: Compliance
Description: Compliances after 8 weeks in each arm or at last visit for early completion. Compliance was calcuated by the percentage of used medication.
Time Frame: 8 weeks for each arm or at last visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of used medication
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
percentage of used medication | 98.4 (3.9) | 97.6 (3.7)
Statistical Analysis 1: Comparison: Once-daily of Ropinirole PR vs Twice-daily of Ropinirole PR; Test type: Superiority or Other; p < 0.05, Sign test; Mean Difference (Net) = 0.8

9. Secondary Outcome: Adverse Events
Description: Patients who have adverse events
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 33 | 28

10. Secondary Outcome: Patients Who Have Global Impression for Improvement
Description: Patients who have global impression for improvement for each dosing.
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: The number of patient who completed the study and answered the questionnaire for global impression.
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 32 | 42

11. Secondary Outcome: Patients Who Have Global Impression for Improvement to Duration of Motor Fluctuation
Description: Patients who have global impression for improvement to duration of motor fluctuation
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: The number of patient who completed the study and answered the questionnaire for global impression to motor fluctuation duration.
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 27 | 38

12. Secondary Outcome: Patients Who Have Global Impression for Improvement to Severity of Motor Fluctuation
Description: Patients who have global impression for improvement to severity of motor fluctuation compared
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: The number of patient who completed the study and answered the questionnaire for global impression to motor fluctuation severity.
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 28 | 34

13. Secondary Outcome: Patients Who Have Global Impression for Improvement to Duration of Dyskinesia
Description: Patients who have global impression for improvement to duration of dyskinesia compared
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: The number of patient who completed the study and answered the questionnaire for global impression to dyskinesia duration.
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 13 | 16

14. Secondary Outcome: Patients Who Have Global Impression for Improvement to Severity of Dyskinesia
Description: Patients who have Global Impression for Improvement to Severity of Dyskinesia compared
Time Frame: After 8 weeks in each arm or at last visit for early completion
Population: The number of patient who completed the study and answered the questionnaire for global impression to dyskinesia severity.
Measure: Number; unit: participants
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Number analyzed (Participants) | 61 | 61
participants | 16 | 15

ADVERSE EVENTS:
Time Frame: 8 weeks for each arm or at last visit
Arm/Group | Once-daily of Ropinirole PR | Twice-daily of Ropinirole PR
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 33/61 | 28/61
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once-daily of Ropinirole PR (N=61) | Twice-daily of Ropinirole PR (N=61)
Nausea (Gastrointestinal disorders) | 9 (9) | 7 (7)
Dizziness (General disorders) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 20 (20) | 19 (19)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3)
Aggravation of vivid dream or REM sleep behavior disorder (Nervous system disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was designed to open-label study. We cannot exclude the psychological effect of each regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No